CLINICAL TRIAL: NCT00541970
Title: Evaluation of the Safety and Immunogenicity of GSK Biologicals' HPV Vaccine 580299 When Administered in Healthy Females Aged 9 - 25 Years Using an Alternative Schedule and an Alternative Dosing as Compared to the Standard Schedule and Dosing
Brief Title: Partially Blind Study to Evaluate Immunogenicity & Safety of GSK Bio's HPV Vaccine 580299 in Healthy Women Aged 9-25 Yrs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 110659
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-08

CONDITIONS: Infections, Papillomavirus
Keywords: viral infections; Human Papillomavirus (HPV) vaccine; safety; vaccine; immunogenicity; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Virus Diseases; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18; halofantrine; Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Cervarix 1/Placebo Group (Experimental): Subjects received 2 doses of the Cervarix vaccine, formulation 1, at Month 0 and Month 2, and 1 dose of placebo at Month 6. The Cervarix vaccine and placebo were administered intramuscularly into the deltoid of the non-dominant arm.
  Interventions: Biological: Cervarix; Drug: Placebo
- Cervarix 1/Placebo/Cervarix 1 Group (Experimental): Subjects received 2 doses of the Cervarix vaccine, formulation 1, at Month 0 and Month 6, and 1 dose of placebo at Month 2. The Cervarix vaccine and placebo were administered intramuscularly into the deltoid of the non-dominant arm.
  Interventions: Biological: Cervarix; Drug: Placebo
- Cervarix 2/Placebo/Cervarix 2 Group (Experimental): Subjects received 2 doses of the Cervarix vaccine, formulation 2, at Month 0 and Month 6, and 1 dose of placebo at Month 2. The Cervarix vaccine and placebo were administered intramuscularly into the deltoid of the non-dominant arm.
  Interventions: Biological: Cervarix; Drug: Placebo
- Cervarix 2 Group (Experimental): Subjects received 3 doses of the Cervarix vaccine, formulation 2, at Month 0, Month 2 and Month 6. The Cervarix vaccine was administered intramuscularly into the deltoid of the non-dominant arm.
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: Cervarix — Intramuscular injection, different dosing /schedule
  Other Names: GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) vaccine 580299
Drug: Placebo — Intramuscular injection, different dosing /schedule
  Arms: Cervarix 1/Placebo Group; Cervarix 1/Placebo/Cervarix 1 Group; Cervarix 2/Placebo/Cervarix 2 Group

SUMMARY:
Human Papillomavirus (HPV) infection has been established as a necessary cause of cervical cancer. GlaxoSmithKline (GSK) Biologicals has developed an HPV vaccine (580299) which targets the 2 most common oncogenic HPV types (HPV-16 and HPV-18), found in approximately 70% of all cervical cancers. In previous trials this vaccine has been found to be efficacious in the prevention of incident and persistent HPV-16/18 infections and associated cytological abnormalities and cervical dysplasia. In this partially-blind study, GSK Biologicals will evaluate the safety and immunogenicity of the HPV vaccine using an alternative schedule and an alternative dosing when administered in healthy young females aged 9 to 25 years, as compared to the standard HPV vaccine. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007. The protocol posting has been updated following a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents can and will comply with the requirements of the protocol should be enrolled in the study.
* A female subject between, and including, 9 and 25 years of age at the time of the first vaccination.
* Written informed consent/assent obtained from the subject prior to enrolment. For subjects above the legal age of consent, written informed consent must be obtained from the subject. For subjects below the legal age of consent, written informed consent from the subject's parents/legally acceptable representative, and written informed assent must be obtained from the subject.
* Healthy subjects as established by medical history and history-oriented clinical examination before entering into the study.
* Subject must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period (up to Month 24).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period (up to Month 24), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. Planned administration/administration of routine vaccines, up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Pregnant or breastfeeding female.
* A woman planning to become pregnant or planning to discontinue contraceptive precautions during the study period, up to two months after the last vaccine dose.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period (up to Month 24).
* Previous administration of components of the investigational vaccine.
* Cancer or autoimmune disease under treatment.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period (up to Month 24).

Ages: 9 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 961 (Actual)
Dates: Start 2007-10-17; Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Québec, Quebec
- Germany (16):
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Rheinstetten, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Nordhausen, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Romanowski B, Schwarz TF, Ferguson LM, Peters K, Dionne M, Schulze K, Ramjattan B, Hillemanns P, Catteau G, Dobbelaere K, Schuind A, Descamps D. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine administered as a 2-dose schedule compared with the licensed 3-dose schedule: results from a randomized study. Hum Vaccin. 2011 Dec;7(12):1374-86. doi: 10.4161/hv.7.12.18322. Epub 2011 Dec 1. PMID 22048171
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Folschweiller N, Behre U, Dionne M, Durando P, Esposito S, Ferguson L, Ferguson M, Hillemanns P, McNeil SA, Peters K, Ramjattan B, Schwarz TF, Supparatpinyo K, Suryakirian PV, Janssens M, Moris P, Decreux A, Poncelet S, Struyf F. Long-term Cross-reactivity Against Nonvaccine Human Papillomavirus Types 31 and 45 After 2- or 3-Dose Schedules of the AS04-Adjuvanted Human HPV-16/18 Vaccine. J Infect Dis. 2019 May 5;219(11):1799-1803. doi: 10.1093/infdis/jiy743. PMID 30715452
- [Derived] Romanowski B, Schwarz TF, Ferguson L, Peters K, Dionne M, Behre U, Schulze K, Hillemanns P, Suryakiran P, Thomas F, Struyf F. Sustained immunogenicity of the HPV-16/18 AS04-adjuvanted vaccine administered as a two-dose schedule in adolescent girls: Five-year clinical data and modeling predictions from a randomized study. Hum Vaccin Immunother. 2016;12(1):20-9. doi: 10.1080/21645515.2015.1065363. Epub 2015 Jul 15. PMID 26176261
- [Derived] Boxus M, Lockman L, Fochesato M, Lorin C, Thomas F, Giannini SL. Antibody avidity measurements in recipients of Cervarix vaccine following a two-dose schedule or a three-dose schedule. Vaccine. 2014 May 30;32(26):3232-6. doi: 10.1016/j.vaccine.2014.04.005. Epub 2014 Apr 13. PMID 24731816
- [Derived] Romanowski B, Schwarz TF, Ferguson LM, Ferguson M, Peters K, Dionne M, Schulze K, Ramjattan B, Hillemanns P, Behre U, Suryakiran P, Thomas F, Struyf F. Immune response to the HPV-16/18 AS04-adjuvanted vaccine administered as a 2-dose or 3-dose schedule up to 4 years after vaccination: results from a randomized study. Hum Vaccin Immunother. 2014;10(5):1155-65. doi: 10.4161/hv.28022. Epub 2014 Feb 27. PMID 24576907
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110659 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included two phases, an active vaccination phase (Months 0-7) followed by a safety follow-up phase (up to the end of the study at Month 60).
Pre-assignment Details: The study was run in an open manner for subjects in the groups receiving the Cervarix vaccine on a 3-dose vaccination schedule. For subjects in the group receiving the Cervarix vaccine on a 2-dose vaccination schedule, the study was run in an observer-blind manner until Month 24, and then in an open manner.
Period: Month 7
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 231 | 228 | 229 | 234
Not Completed | 9 | 13 | 11 | 5
Not completed — Protocol Violation | 9 | 13 | 11 | 5
Period: Month 12
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 228 | 219 | 219 | 223
Not Completed | 12 | 22 | 21 | 16
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 12 | 21 | 20 | 15
Period: Month 18
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 226 | 217 | 215 | 222
Not Completed | 14 | 24 | 25 | 17
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 14 | 23 | 24 | 16
Period: Month 24
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 211 | 209 | 208 | 217
Not Completed | 29 | 32 | 32 | 22
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 29 | 31 | 31 | 21
Period: Month 36
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 179 | 175 | 174 | 179
Not Completed | 61 | 66 | 66 | 60
Not completed — Protocol Violation | 61 | 66 | 66 | 60
Period: Month 48
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 169 | 168 | 167 | 164
Not Completed | 71 | 73 | 73 | 75
Not completed — Withdrawal by Subject | 2 | 4 | 4 | 2
Not completed — Other | 3 | 1 | 1 | 0
Not completed — Lost to Follow-up | 66 | 68 | 68 | 73
Period: Month 60
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Started | 240 | 241 | 240 | 239
Completed | 162 | 164 | 158 | 167
Not Completed | 78 | 77 | 82 | 72
Not completed — Protocol Violation | 78 | 77 | 82 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group | Total
Number analyzed (Participants) | 240 | 241 | 240 | 239 | 960
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.1 (4.30) | 17.2 (4.30) | 17.3 (4.25) | 17.2 (4.38) | 17.2 (4.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 241 | 240 | 239 | 960
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Titers of Anti-Papillomavirus 16 (Anti-HPV-16) and Anti-human Papillomavirus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed in Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: One month after vaccination with the last dose of the Cervarix vaccine (Cervarix 1/Placebo Group: Month 3; Other groups: Month 7).
Population: The analysis was performed on the According-to-Protocol cohort for Immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 224 | 206 | 204 | 208
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 224 | 204 | 204 | 208
  Anti-HPV-16 | 5844.6 [5259.6 to 6494.7] | 10500.9 [9356.9 to 11784.8] | 7741.6 [6868.2 to 8726.1] | 13045.3 [11211.4 to 15179.2]
  Anti-HPV-18: number analyzed (Participants) | 223 | 206 | 204 | 208
  Anti-HPV-18 | 3543.2 [3126.6 to 4015.3] | 5997.5 [5310.9 to 6772.8] | 4811.4 [4282.7 to 5405.3] | 5087.1 [4460.2 to 5802.1]

2. Primary Outcome: Number of Subjects With Report of Any, and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the solicited local symptom irrespective of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling larger than (>) 50 millimeters (mm).
Time Frame: Within 7 days (Day 0-6) after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented. Analysis for this outcome was done on subjects with available results for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 238 | 239 | 238 | 238
Participants
  Any Pain | 222 | 225 | 222 | 225
  Grade 3 Pain | 18 | 27 | 26 | 35
  Any Redness | 109 | 112 | 123 | 145
  Redness > 50 mm | 3 | 4 | 1 | 3
  Any Swelling | 92 | 88 | 83 | 118
  Swelling > 50 mm | 4 | 3 | 1 | 5

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever (defined as axillary temperature equal or above (≥) 37.5 degrees Celsius (°C), gastrointestinal symptoms, which included nausea, vomiting, diarrhoea and/or abdominal pain, headache, myalgia, rash and urticaria. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature ≥ 39 °C. Grade 3 urticaria = urticaria distributed on at least 4 body areas. Related symptom = symptom assessed by the investigator to be causally related to vaccination.
Time Frame: Within 7 days (Day 0-6) after vaccination.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 238 | 239 | 238 | 238
Participants
  Any Arthralgia | 45 | 57 | 39 | 43
  Related Arthralgia | 39 | 43 | 35 | 35
  Grade 3 Arthralgia | 0 | 3 | 4 | 3
  Any Fatigue | 100 | 109 | 104 | 107
  Related Fatigue | 76 | 82 | 87 | 83
  Grade 3 Fatigue | 11 | 4 | 5 | 8
  Any Fever (Axillary Temperature >= 37.5°C) | 23 | 20 | 22 | 39
  Related Fever | 18 | 15 | 16 | 27
  Grade 3 Fever (Axillary Temperature >= 39.0°C) | 1 | 0 | 1 | 0
  Any Gastrointestinal Symptoms | 48 | 48 | 36 | 68
  Related Gastrointestinal Symptoms | 36 | 43 | 27 | 50
  Grade 3 Gastrointestinal Symptoms | 3 | 7 | 2 | 7
  Any Headache | 101 | 116 | 112 | 125
  Related Headache | 79 | 81 | 91 | 95
  Grade 3 Headache | 9 | 9 | 7 | 12
  Any Myalgia | 79 | 109 | 98 | 99
  Related Myalgia | 62 | 87 | 75 | 77
  Grade 3 Myalgia | 3 | 9 | 6 | 7
  Any Rash | 12 | 12 | 10 | 15
  Related Rash | 8 | 9 | 8 | 9
  Grade 3 Rash | 0 | 0 | 1 | 1
  Any Urticaria | 2 | 4 | 4 | 5
  Related Urticaria | 1 | 3 | 4 | 3
  Grade 3 Urticaria | 0 | 0 | 1 | 0

4. Secondary Outcome: Titers of Anti-Papillomavirus 16 (Anti-HPV-16) and Anti-human Papillomavirus 18 (Anti-HPV-18) Antibodies .
Description: Titers are given as Geometric Mean Titers (GMTs) expressed in Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). The analysis was performed on the subjects who were administered a 2-dose vaccination schedule.
Time Frame: At Month 3, 1 month after the second dose of vaccine or placebo
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group
Number analyzed (Participants) | 224 | 206 | 203
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 224 | 204 | 203
  Anti-HPV-16 | 5844.6 [5259.6 to 6494.7] | 397.9 [337.4 to 469.2] | 266.4 [227.2 to 312.4]
  Anti-HPV-18: number analyzed (Participants) | 223 | 206 | 203
  Anti-HPV-18 | 3543.2 [3126.6 to 4015.3] | 228.3 [196.7 to 265.0] | 181.9 [156.8 to 211.1]

5. Secondary Outcome: Titers of Anti-Papillomavirus 16 (Anti-HPV-16) and Anti-human Papillomavirus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed in Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). Groups were stratified into 3 age strata: 9-14, 15-19 and 20-25 years of age at the time of first vaccination. The 15-19 years age stratum in the group receiving the Cervarix vaccine on a 3-dose vaccination schedule was considered an active comparator.
Time Frame: At Month 7, 1 month after the last dose of vaccine or placebo.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 221 | 206 | 204 | 208
EL.U/mL
  9-14 years, Anti-HPV-16: number analyzed (Participants) | 76 | 62 | 69 | 75
  9-14 years, Anti-HPV-16 | 2003.9 [1635.7 to 2455.0] | 15028.4 [12611.3 to 17908.6] | 11058.6 [9273.8 to 13186.7] | 22066.3 [18140.7 to 26841.2]
  15-19 years, Anti-HPV-16: number analyzed (Participants) | 72 | 74 | 70 | 66
  15-19 years, Anti-HPV-16 | 1168.5 [957.4 to 1426.2] | 10818.7 [8979.8 to 13034.2] | 7869.6 [6488.9 to 9543.9] | 12817.4 [9723.2 to 16896.2]
  20-25 years, Anti-HPV-16: number analyzed (Participants) | 73 | 68 | 65 | 67
  20-25 years, Anti-HPV-16 | 1371.2 [1092.2 to 1721.6] | 7331.4 [5965.2 to 9010.4] | 5209.2 [4166.5 to 6512.7] | 7370.0 [5673.6 to 9573.6]
  9-14 years, Anti-HPV-18: number analyzed (Participants) | 76 | 64 | 69 | 75
  9-14 years, Anti-HPV-18 | 1134.3 [922.8 to 1394.3] | 8085.8 [6654.5 to 9825.0] | 5630.7 [4772.1 to 6643.7] | 7192.9 [5952.6 to 8691.6]
  15-19 years, Anti-HPV-18: number analyzed (Participants) | 72 | 74 | 69 | 66
  15-19 years, Anti-HPV-18 | 719.8 [571.2 to 907.0] | 6170.1 [5046.8 to 7543.5] | 5039.3 [4283.4 to 5928.5] | 4907.0 [3780.8 to 6368.7]
  20-25 years, Anti-HPV-18: number analyzed (Participants) | 72 | 68 | 66 | 67
  20-25 years, Anti-HPV-18 | 656.5 [514.6 to 837.5] | 4389.6 [3525.6 to 5465.4] | 3889.2 [2980.9 to 5074.3] | 3576.8 [2886.5 to 4432.2]

6. Secondary Outcome: Titers of Anti-Papillomavirus 16 (Anti-HPV-16) and Anti-human Papillomavirus 18 (Anti-HPV-18) Antibodies
Description: as for outcome 1
Time Frame: At Month 12, at Month 18, at Month 24, at Month 36, and at Month 48 during the safety follow-up phase.
Population: The analysis was performed on the According-to-Protocol cohort for Immunogenicity, which included all evaluable subjects eligible for whom immunogenicity data were available, and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 216 | 198 | 195 | 198
EL.U/mL
  Anti-HPV-16 at Month 12: number analyzed (Participants) | 216 | 191 | 195 | 198
  Anti-HPV-16 at Month 12 | 1064.7 [937.5 to 1209.1] | 3256.0 [2918.8 to 3632.1] | 2438.7 [2167.2 to 2744.2] | 4726.7 [4036.8 to 5534.6]
  Anti-HPV-16 at Month 18: number analyzed (Participants) | 212 | 196 | 194 | 197
  Anti-HPV-16 at Month 18 | 968.1 [845.2 to 1109.0] | 2229.4 [1983.2 to 2506.2] | 1659.1 [1466.9 to 1876.4] | 3185.1 [2735.1 to 3709.2]
  Anti-HPV-16 at Month 24: number analyzed (Participants) | 199 | 184 | 186 | 190
  Anti-HPV-16 at Month 24 | 821.2 [718.5 to 938.5] | 1756.4 [1556.6 to 1981.9] | 1285.1 [1139.6 to 1449.2] | 2425.9 [2071.1 to 2841.5]
  Anti-HPV-16 at Month 36: number analyzed (Participants) | 166 | 158 | 162 | 153
  Anti-HPV-16 at Month 36 | 688.3 [592.2 to 799.9] | 1462.2 [1288.8 to 1658.8] | 1094.0 [961.1 to 1245.1] | 2195.4 [1850.8 to 2604.1]
  Anti-HPV-16 at Month 48: number analyzed (Participants) | 160 | 151 | 157 | 148
  Anti-HPV-16 at Month 48 | 649.5 [556.0 to 758.8] | 1261.2 [1106.4 to 1437.7] | 953.5 [835.5 to 1088.2] | 1892.3 [1594.2 to 2246.0]
  Anti-HPV-18 at Month 12: number analyzed (Participants) | 215 | 193 | 194 | 198
  Anti-HPV-18 at Month 12 | 472.9 [410.5 to 544.8] | 1760.1 [1531.5 to 2022.8] | 1426.2 [1250.8 to 1626.1] | 1714.5 [1469.7 to 2000.0]
  Anti-HPV-18 at Month 18: number analyzed (Participants) | 211 | 198 | 193 | 197
  Anti-HPV-18 at Month 18 | 389.2 [338.7 to 447.2] | 1025.2 [889.0 to 1182.2] | 883.1 [774.7 to 1006.8] | 1096.6 [939.4 to 1280.1]
  Anti-HPV-18 at Month 24: number analyzed (Participants) | 198 | 186 | 185 | 190
  Anti-HPV-18 at Month 24 | 345.9 [299.3 to 399.8] | 818.2 [706.5 to 947.5] | 674.6 [591.8 to 769.0] | 866.8 [741.2 to 1013.6]
  Anti-HPV-18 at Month 36: number analyzed (Participants) | 166 | 160 | 162 | 153
  Anti-HPV-18 at Month 36 | 302.2 [254.9 to 358.2] | 712.8 [605.4 to 839.3] | 617.9 [532.3 to 717.2] | 874.2 [734.9 to 1040.0]
  Anti-HPV-18 at Month 48: number analyzed (Participants) | 160 | 153 | 157 | 148
  Anti-HPV-18 at Month 48 | 260.4 [218.5 to 310.2] | 626.3 [531.0 to 738.7] | 517.0 [446.2 to 599.1] | 723.2 [607.2 to 861.4]

7. Secondary Outcome: Titers of Anti-Papillomavirus 16 (Anti-HPV-16) and Anti-human Papillomavirus 18 (Anti-HPV-18) Antibodies
Description: as for outcome 1
Time Frame: At Month 7, 1 month after the last dose of vaccine or placebo.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 221 | 206 | 204 | 208
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 221 | 204 | 204 | 208
  Anti-HPV-16 | 1677.5 [1677.5 to 1677.5] | 11784.8 [11784.8 to 11784.8] | 8726.1 [8726.1 to 8726.1] | 15179.2 [15179.2 to 15179.2]
  Anti-HPV-18: number analyzed (Participants) | 220 | 206 | 204 | 208
  Anti-HPV-18 | 817.3 [715.6 to 933.4] | 5997.5 [5310.9 to 6772.8] | 4811.4 [4282.7 to 5405.3] | 5087.1 [4460.2 to 5802.1]

8. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents BAS results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 223 | 221 | 221 | 225
Participants
  BAS, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 222 | 219 | 218 | 220
  BAS, PRE NORMAL, M7 NORMAL | 219 | 214 | 208 | 214
  BAS, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 222 | 219 | 218 | 220
  BAS, PRE NORMAL, M7 BELOW | 0 | 0 | 0 | 0
  BAS, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 222 | 219 | 218 | 220
  BAS, PRE NORMAL, M7 ABOVE | 2 | 3 | 6 | 3
  BAS, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 222 | 219 | 218 | 220
  BAS, PRE NORMAL, M7 MISSING | 1 | 2 | 4 | 3
  BAS, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 0 | 0 | 1 | 1
  BAS, PRE BELOW, M7 NORMAL | 0 | 0 | 1 | 0
  BAS, PRE BELOW, M7 BELOW: number analyzed (Participants) | 0 | 0 | 1 | 1
  BAS, PRE BELOW, M7 BELOW | 0 | 0 | 0 | 1
  BAS, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 0 | 0 | 1 | 1
  BAS, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  BAS, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 1 | 2 | 2 | 4
  BAS, PRE ABOVE, M7 NORMAL | 1 | 2 | 2 | 4
  BAS, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 1 | 2 | 2 | 4
  BAS, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  BAS, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 1 | 2 | 2 | 4
  BAS, PRE ABOVE, M7 ABOVE | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range.This outcome presents CREA results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 226 | 225 | 228 | 229
Participants
  CREA, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 215 | 211 | 215 | 218
  CREA, PRE NORMAL, M7 NORMAL | 202 | 200 | 210 | 206
  CREA, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 215 | 211 | 215 | 218
  CREA, PRE NORMAL, M7 BELOW | 7 | 4 | 3 | 6
  CREA, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 215 | 211 | 215 | 218
  CREA, PRE NORMAL, M7 ABOVE | 5 | 7 | 1 | 4
  CREA, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 215 | 211 | 215 | 218
  CREA, PRE NORMAL, M7 MISSING | 1 | 0 | 1 | 2
  CREA, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 8 | 7 | 7 | 6
  CREA, PRE BELOW, M7 NORMAL | 6 | 3 | 3 | 2
  CREA, PRE BELOW, M7 BELOW: number analyzed (Participants) | 8 | 7 | 7 | 6
  CREA, PRE BELOW, M7 BELOW | 2 | 4 | 4 | 3
  CREA, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 8 | 7 | 7 | 6
  CREA, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  CREA, PRE BELOW, M7 MISSING: number analyzed (Participants) | 8 | 7 | 7 | 6
  CREA, PRE BELOW, M7 MISSING | 0 | 0 | 0 | 1
  CREA, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 3 | 7 | 6 | 5
  CREA, PRE ABOVE, M7 NORMAL | 2 | 4 | 4 | 2
  CREA, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 3 | 7 | 6 | 5
  CREA, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  CREA, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 3 | 7 | 6 | 5
  CREA, PRE ABOVE, M7 ABOVE | 1 | 3 | 2 | 3

10. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents EOS results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 226 | 223 | 223 | 226
Participants
  EOS, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 209 | 214 | 212 | 214
  EOS, PRE NORMAL, M7 NORMAL | 203 | 207 | 200 | 205
  EOS, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 226 | 214 | 212 | 214
  EOS, PRE NORMAL, M7 BELOW | 0 | 0 | 0 | 0
  EOS, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 209 | 214 | 212 | 214
  EOS, PRE NORMAL, M7 ABOVE | 5 | 6 | 8 | 6
  EOS, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 209 | 214 | 212 | 214
  EOS, PRE NORMAL, M7 MISSING | 1 | 1 | 4 | 3
  EOS, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 1 | 2 | 1 | 0
  EOS, PRE BELOW, M7 NORMAL | 0 | 1 | 0 | 0
  EOS, PRE BELOW, M7 BELOW: number analyzed (Participants) | 1 | 2 | 1 | 0
  EOS, PRE BELOW, M7 BELOW | 0 | 1 | 1 | 0
  EOS, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 1 | 2 | 1 | 0
  EOS, PRE BELOW, M7 ABOVE | 1 | 0 | 0 | 0
  EOS, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 16 | 7 | 10 | 12
  EOS, PRE ABOVE, M7 NORMAL | 8 | 3 | 3 | 7
  EOS, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 16 | 7 | 10 | 12
  EOS, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  EOS, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 16 | 7 | 10 | 12
  EOS, PRE ABOVE, M7 ABOVE | 8 | 3 | 7 | 5
  EOS, PRE ABOVE, M7 MISSING: number analyzed (Participants) | 16 | 7 | 10 | 12
  EOS, PRE ABOVE, M7 MISSING | 0 | 1 | 0 | 0

11. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents Hct results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 229 | 228 | 227 | 233
Participants
  Hct, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 215 | 208 | 208 | 217
  Hct, PRE NORMAL, M7 NORMAL | 196 | 193 | 189 | 208
  Hct, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 215 | 208 | 208 | 217
  Hct, PRE NORMAL, M7 BELOW | 6 | 5 | 8 | 2
  Hct, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 215 | 208 | 208 | 217
  Hct, PRE NORMAL, M7 ABOVE | 11 | 8 | 7 | 6
  Hct, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 215 | 208 | 208 | 217
  Hct, PRE NORMAL, M7 MISSING | 2 | 2 | 4 | 1
  Hct, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 6 | 7 | 7 | 3
  Hct, PRE BELOW, M7 NORMAL | 3 | 5 | 4 | 2
  Hct, PRE BELOW, M7 BELOW: number analyzed (Participants) | 6 | 7 | 7 | 3
  Hct, PRE BELOW, M7 BELOW | 3 | 2 | 3 | 1
  Hct, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 6 | 7 | 7 | 3
  Hct, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  Hct, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 8 | 13 | 12 | 13
  Hct, PRE ABOVE, M7 NORMAL | 7 | 8 | 10 | 7
  Hct, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 8 | 13 | 12 | 13
  Hct, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  Hct, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 8 | 13 | 12 | 13
  Hct, PRE ABOVE, M7 ABOVE | 1 | 5 | 2 | 6

12. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents ALT results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 229 | 227 | 229 | 233
Participants
  ALT, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 215 | 219 | 225 | 218
  ALT, PRE NORMAL, M7 NORMAL | 211 | 211 | 213 | 209
  ALT, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 215 | 219 | 225 | 218
  ALT, PRE NORMAL, M7 BELOW | 3 | 2 | 4 | 4
  ALT, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 215 | 219 | 225 | 218
  ALT, PRE NORMAL, M7 ABOVE | 1 | 6 | 7 | 5
  ALT, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 215 | 219 | 225 | 218
  ALT, PRE NORMAL, M7 MISSING | 0 | 0 | 1 | 0
  ALT, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 1 | 3 | 1 | 4
  ALT, PRE BELOW, M7 NORMAL | 0 | 2 | 0 | 2
  ALT, PRE BELOW, M7 BELOW: number analyzed (Participants) | 1 | 3 | 1 | 4
  ALT, PRE BELOW, M7 BELOW | 1 | 1 | 1 | 2
  ALT, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 1 | 3 | 1 | 4
  ALT, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  ALT, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 13 | 5 | 3 | 11
  ALT, PRE ABOVE, M7 NORMAL | 9 | 4 | 1 | 7
  ALT, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 13 | 5 | 3 | 11
  ALT, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  ALT, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 13 | 5 | 3 | 11
  ALT, PRE ABOVE, M7 ABOVE | 4 | 1 | 2 | 3
  ALT, PRE ABOVE, M7 MISSING: number analyzed (Participants) | 13 | 5 | 3 | 11
  ALT, PRE ABOVE, M7 MISSING | 0 | 0 | 0 | 1

13. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents LYM results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 226 | 223 | 223 | 227
Participants
  LYM, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 211 | 211 | 204 | 213
  LYM, PRE NORMAL, M7 NORMAL | 201 | 202 | 192 | 202
  LYM, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 211 | 211 | 204 | 213
  LYM, PRE NORMAL, M7 BELOW | 3 | 0 | 3 | 1
  LYM, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 211 | 211 | 204 | 213
  LYM, PRE NORMAL, M7 ABOVE | 6 | 7 | 5 | 7
  LYM, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 211 | 211 | 204 | 213
  LYM, PRE NORMAL, M7 MISSING | 1 | 2 | 4 | 3
  LYM, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 6 | 3 | 5 | 5
  LYM, PRE BELOW, M7 NORMAL | 4 | 3 | 3 | 1
  LYM, PRE BELOW, M7 BELOW: number analyzed (Participants) | 6 | 3 | 5 | 5
  LYM, PRE BELOW, M7 BELOW | 2 | 0 | 2 | 2
  LYM, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 6 | 3 | 5 | 5
  LYM, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 2
  LYM, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 9 | 9 | 14 | 9
  LYM, PRE ABOVE, M7 NORMAL | 5 | 7 | 8 | 5
  LYM, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 9 | 9 | 14 | 9
  LYM, PRE ABOVE, M7 BELOW | 0 | 0 | 1 | 0
  LYM, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 9 | 9 | 14 | 9
  LYM, PRE ABOVE, M7 ABOVE | 4 | 2 | 5 | 4

14. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents MON results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 226 | 223 | 223 | 227
Participants
  MON, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 217 | 211 | 211 | 219
  MON, PRE NORMAL, M7 NORMAL | 212 | 202 | 197 | 208
  MON, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 217 | 211 | 211 | 219
  MON, PRE NORMAL, M7 BELOW | 0 | 1 | 2 | 2
  MON, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 217 | 211 | 211 | 219
  MON, PRE NORMAL, M7 ABOVE | 4 | 6 | 9 | 6
  MON, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 217 | 211 | 211 | 219
  MON, PRE NORMAL, M7 MISSING | 1 | 2 | 3 | 3
  MON, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 3 | 2 | 0 | 2
  MON, PRE BELOW, M7 NORMAL | 1 | 1 | 0 | 2
  MON, PRE BELOW, M7 BELOW: number analyzed (Participants) | 3 | 2 | 0 | 2
  MON, PRE BELOW, M7 BELOW | 2 | 1 | 0 | 0
  MON, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 3 | 2 | 0 | 2
  MON, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  MON, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 6 | 10 | 12 | 6
  MON, PRE ABOVE, M7 NORMAL | 5 | 6 | 6 | 4
  MON, PRE ABOVE], M7 BELOW: number analyzed (Participants) | 6 | 10 | 12 | 6
  MON, PRE ABOVE], M7 BELOW | 0 | 0 | 0 | 0
  MON, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 6 | 10 | 12 | 6
  MON, PRE ABOVE, M7 ABOVE | 1 | 4 | 5 | 2
  MON, PRE ABOVE, M7 MISSING: number analyzed (Participants) | 6 | 10 | 12 | 6
  MON, PRE ABOVE, M7 MISSING | 0 | 0 | 1 | 0

15. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents NEU results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 224 | 223 | 223 | 226
Participants
  NEU, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 206 | 207 | 202 | 204
  NEU, PRE NORMAL, M7 NORMAL | 184 | 188 | 185 | 186
  NEU, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 206 | 207 | 202 | 204
  NEU, PRE NORMAL, M7 BELOW | 16 | 16 | 9 | 9
  NEU, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 206 | 207 | 202 | 204
  NEU, PRE NORMAL, M7 ABOVE | 5 | 1 | 1 | 3
  NEU, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 206 | 207 | 202 | 204
  NEU, PRE NORMAL, M7 MISSING | 1 | 2 | 7 | 6
  NEU, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 11 | 11 | 16 | 19
  NEU, PRE BELOW, M7 NORMAL | 8 | 6 | 9 | 15
  NEU, PRE BELOW, M7 BELOW: number analyzed (Participants) | 11 | 11 | 16 | 19
  NEU, PRE BELOW, M7 BELOW | 2 | 4 | 7 | 3
  NEU, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 11 | 11 | 16 | 19
  NEU, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  NEU, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 7 | 5 | 5 | 3
  NEU, PRE ABOVE, M7 NORMAL | 6 | 5 | 5 | 1
  NEU, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 7 | 5 | 5 | 3
  NEU, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 2
  NEU, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 7 | 5 | 5 | 3
  NEU, PRE ABOVE, M7 ABOVE | 1 | 0 | 0 | 0
  NEU, PRE BELOW, M7 MISSING: number analyzed (Participants) | 11 | 11 | 16 | 19
  NEU, PRE BELOW, M7 MISSING | 1 | 1 | 0 | 1

16. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents RBC results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 229 | 228 | 228 | 233
Participants
  RBC, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 214 | 215 | 204 | 225
  RBC, PRE NORMAL, M7 NORMAL | 204 | 204 | 196 | 213
  RBC, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 214 | 215 | 204 | 225
  RBC, PRE NORMAL, M7 BELOW | 7 | 7 | 2 | 7
  RBC, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 214 | 215 | 204 | 225
  RBC, PRE NORMAL, M7 ABOVE | 2 | 3 | 2 | 3
  RBC, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 214 | 215 | 204 | 225
  RBC, PRE NORMAL, M7 MISSING | 1 | 1 | 4 | 2
  RBC, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 6 | 6 | 12 | 4
  RBC, PRE BELOW, M7 NORMAL | 4 | 3 | 2 | 1
  RBC, PRE BELOW, M7 BELOW: number analyzed (Participants) | 6 | 6 | 12 | 4
  RBC, PRE BELOW, M7 BELOW | 2 | 3 | 10 | 3
  RBC, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 6 | 6 | 12 | 4
  RBC, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  RBC, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 9 | 7 | 12 | 4
  RBC, PRE ABOVE, M7 NORMAL | 5 | 4 | 6 | 3
  RBC, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 9 | 7 | 12 | 4
  RBC, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  RBC, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 9 | 7 | 12 | 4
  RBC, PRE ABOVE, M7 ABOVE | 4 | 3 | 6 | 1

17. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents WBC results.
Time Frame: At Month 7 (M7)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented, on subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 229 | 228 | 229 | 233
Participants
  WBC, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 207 | 213 | 211 | 225
  WBC, PRE NORMAL, M7 NORMAL | 197 | 199 | 194 | 212
  WBC, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 207 | 213 | 211 | 225
  WBC, PRE NORMAL, M7 BELOW | 4 | 9 | 5 | 9
  WBC, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 207 | 213 | 211 | 225
  WBC, PRE NORMAL, M7 ABOVE | 5 | 4 | 8 | 3
  WBC, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 207 | 213 | 211 | 225
  WBC, PRE NORMAL, M7 MISSING | 1 | 1 | 4 | 1
  WBC, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 8 | 9 | 6 | 4
  WBC, PRE BELOW, M7 NORMAL | 4 | 5 | 3 | 3
  WBC, PRE BELOW, M7 BELOW: number analyzed (Participants) | 8 | 9 | 6 | 4
  WBC, PRE BELOW, M7 BELOW | 4 | 4 | 3 | 1
  WBC, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 8 | 9 | 6 | 4
  WBC, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  WBC, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 14 | 6 | 12 | 4
  WBC, PRE ABOVE, M7 NORMAL | 10 | 4 | 9 | 4
  WBC, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 14 | 6 | 12 | 4
  WBC, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  WBC, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 14 | 6 | 12 | 4
  WBC, PRE ABOVE, M7 ABOVE | 4 | 2 | 3 | 0

18. Secondary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Biochemical and Haematological Laboratory Parameters Assessed.
Description: Assessed parameters were alanine aminotransferase (ALT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocritis (Hct), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). Subjects were categorized according to their results at pre-vaccination at Month 0 (PRE) which were normal, above normal or below the normal range. Per parameter and range, it was assessed whether laboratory values of the subjects were normal, above normal or below the normal range. This outcome presents PLA results.
Time Frame: At Month 7 (M7)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 226 | 227 | 228 | 232
Participants
  PLA, PRE NORMAL, M7 NORMAL: number analyzed (Participants) | 211 | 210 | 215 | 221
  PLA, PRE NORMAL, M7 NORMAL | 204 | 204 | 206 | 218
  PLA, PRE NORMAL, M7 BELOW: number analyzed (Participants) | 211 | 210 | 215 | 221
  PLA, PRE NORMAL, M7 BELOW | 1 | 2 | 3 | 0
  PLA, PRE NORMAL, M7 ABOVE: number analyzed (Participants) | 211 | 210 | 215 | 221
  PLA, PRE NORMAL, M7 ABOVE | 5 | 2 | 2 | 1
  PLA, PRE NORMAL, M7 MISSING: number analyzed (Participants) | 211 | 210 | 215 | 221
  PLA, PRE NORMAL, M7 MISSING | 1 | 2 | 4 | 2
  PLA, PRE BELOW, M7 NORMAL: number analyzed (Participants) | 0 | 3 | 0 | 3
  PLA, PRE BELOW, M7 NORMAL | 0 | 0 | 0 | 1
  PLA, PRE BELOW, M7 BELOW: number analyzed (Participants) | 0 | 3 | 0 | 3
  PLA, PRE BELOW, M7 BELOW | 0 | 3 | 0 | 2
  PLA, PRE BELOW, M7 ABOVE: number analyzed (Participants) | 0 | 3 | 0 | 3
  PLA, PRE BELOW, M7 ABOVE | 0 | 0 | 0 | 0
  PLA, PRE ABOVE, M7 NORMAL: number analyzed (Participants) | 15 | 14 | 13 | 8
  PLA, PRE ABOVE, M7 NORMAL | 9 | 11 | 8 | 4
  PLA, PRE ABOVE, M7 BELOW: number analyzed (Participants) | 15 | 14 | 13 | 8
  PLA, PRE ABOVE, M7 BELOW | 0 | 0 | 0 | 0
  PLA, PRE ABOVE, M7 ABOVE: number analyzed (Participants) | 15 | 14 | 13 | 8
  PLA, PRE ABOVE, M7 ABOVE | 6 | 3 | 5 | 4

19. Secondary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus 16 (HPV-16) and Human Papillomavirus 18 (HPV-18)
Description: Seroconversion was defined as the appearance of antibodies (i.e.titers greater than or equal to (≥) cut-off value) in the serum of subjects seronegative before vaccination. Assay cut-off was defined as ≥ 8 ELISA units per milliliter (EL.U/mL) for HPV-16, and 7 EL.U/mL for HPV-18. Seronegative subjects are subjects who had an antibody concentration below cut-off value. Cut-off values were 8 EL.U/mL for antibody concentrations against HPV-16, and 7 EL.U/mL for antibody concentrations against HPV-18.
Time Frame: At Month 12, at Month 18, at Month 24, at Month 36, and at Month 48 during the safety follow-up phase.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 216 | 198 | 195 | 198
Participants
  Anti-HPV-16 at Month 12: number analyzed (Participants) | 216 | 191 | 195 | 198
  Anti-HPV-16 at Month 12 | 194 | 162 | 172 | 169
  Anti-HPV-16 at Month 18: number analyzed (Participants) | 212 | 196 | 194 | 197
  Anti-HPV-16 at Month 18 | 192 | 166 | 172 | 168
  Anti-HPV-16 at Month 24: number analyzed (Participants) | 199 | 184 | 186 | 190
  Anti-HPV-16 at Month 24 | 185 | 155 | 165 | 162
  Anti-HPV-16 at Month 36: number analyzed (Participants) | 166 | 158 | 162 | 153
  Anti-HPV-16 at Month 36 | 156 | 135 | 146 | 135
  Anti-HPV-16 at Month 48: number analyzed (Participants) | 160 | 151 | 157 | 148
  Anti-HPV-16 at Month 48 | 149 | 130 | 139 | 129
  Anti-HPV-18 at Month 12: number analyzed (Participants) | 215 | 193 | 194 | 198
  Anti-HPV-18 at Month 12 | 187 | 173 | 166 | 173
  Anti-HPV-18 at Month 18: number analyzed (Participants) | 211 | 198 | 193 | 197
  Anti-HPV-18 at Month 18 | 184 | 177 | 166 | 173
  Anti-HPV-18 at Month 24: number analyzed (Participants) | 198 | 186 | 185 | 190
  Anti-HPV-18 at Month 24 | 173 | 165 | 159 | 166
  Anti-HPV-18 at Month 36: number analyzed (Participants) | 166 | 160 | 162 | 153
  Anti-HPV-18 at Month 36 | 144 | 145 | 139 | 132
  Anti-HPV-18 at Month 48: number analyzed (Participants) | 160 | 153 | 157 | 148
  Anti-HPV-18 at Month 48 | 138 | 139 | 135 | 129

20. Secondary Outcome: Titers of Anti-Papillomavirus 16 (Anti-HPV-16) and Anti-human Papillomavirus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed in Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). The assay cut-off for Month 60 was defined as ≥ 19 ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 60 of the safety follow-up phase
Population: The analysis was performed on the ATP cohort for Immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 137 | 134 | 131 | 146
EL.U/mL
  Anti-HPV-16 at Month 60: number analyzed (Participants) | 137 | 132 | 131 | 146
  Anti-HPV-16 at Month 60 | 658.0 [560.4 to 772.5] | 1254.0 [1088.5 to 1444.8] | 976.1 [846.1 to 1126.1] | 1858.5 [1586.2 to 2177.6]
  Anti-HPV-18 at Month 60 | 269.4 [223.0 to 325.5] | 622.2 [519.0 to 745.9] | 557.9 [473.7 to 657.0] | 745.3 [629.3 to 882.7]

21. Secondary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus 16 (HPV-16) and Human Papillomavirus 18 (HPV-18)
Description: Seroconversion was defined as the appearance of antibodies (i.e. titers greater than or equal to (≥) cut-off value) in the serum of subjects seronegative before vaccination. Assay cut-off was defined as ≥ 19 ELISA units per milliliter (EL.U/mL). Seronegative subjects are subjects who had an antibody concentration below cut-off value.
Time Frame: At Month 60 of the safety follow-up phase
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 130 | 122 | 119 | 127
Participants
  Anti-HPV-16 at Month 60: number analyzed (Participants) | 130 | 114 | 119 | 127
  Anti-HPV-16 at Month 60 | 130 | 114 | 119 | 127
  Anti-HPV-18 at Month 60: number analyzed (Participants) | 117 | 122 | 116 | 125
  Anti-HPV-18 at Month 60 | 116 | 122 | 116 | 125

22. Secondary Outcome: Number of Subjects With Pregnancy Outcomes.
Description: Pregnancy outcomes were ectopic pregnancy, elective termination with no apparent congenital anomaly (ACA), elective termination with congenital anomaly (CA), lost to follow up, pregnancy ongoing, spontaneous abortion with no ACA and live infant with no ACA.
Time Frame: From Month 0 to Month 48.
Population: The analysis was performed on pregnant subjects in the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 23 | 16 | 24 | 20
Participants
  Ectopic pregnancy | 1 | 0 | 0 | 0
  Elective termination with NO ACA | 5 | 3 | 3 | 5
  Elective termination with CA | 0 | 0 | 1 | 0
  Live infant with NO ACA | 15 | 12 | 15 | 12
  Lost to follow up | 1 | 0 | 0 | 0
  Pregnancy ongoing | 0 | 1 | 2 | 2
  Spontaneous abortion with NO ACA | 1 | 0 | 3 | 1

23. Secondary Outcome: Number of Subjects With Pregnancy Outcomes.
Description: as for outcome 22
Time Frame: Throughout the study period, from Month 0 to Month 60.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 32 | 23 | 30 | 26
Participants
  Ectopic pregnancy | 1 | 0 | 0 | 1
  Elective termination NO apparent congenital anom. | 5 | 6 | 4 | 6
  Elective termination congenital anomaly | 0 | 0 | 1 | 0
  Live infant NO apparent congenital anomaly | 22 | 16 | 22 | 18
  Lost to follow up | 1 | 0 | 0 | 0
  Molar pregnancy | 1 | 0 | 0 | 0
  Spontaneous abortion NO apparent congenital anom. | 2 | 1 | 3 | 1

24. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event (AE) is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Grade 3 = an event that prevented normal activity. Related = an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 30 days (Day 0-29) after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants
  Any unsolicited AE(s) | 83 | 85 | 76 | 107
  Grade 3 unsolicited AE(s) | 11 | 8 | 6 | 14
  Related unsolicited AE(s) | 26 | 20 | 16 | 27

25. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs).
Description: MSCs were defined as: AEs prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that were not related to common diseases. The following did not require reporting as long as they were not considered SAEs and occurred more than 30 days after each vaccination: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities, injury, visits for routine physical examination or visits for vaccination.
Time Frame: From Month 0 to Month 7.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 40 | 48 | 45 | 42

26. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs).
Description: as for outcome 25
Time Frame: From Month 0 to Month 48.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 79 | 94 | 88 | 82

27. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs).
Description: as for outcome 25
Time Frame: Throughout the study period, from Month 0 to Month 60.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 85 | 97 | 92 | 89

28. Secondary Outcome: Number of Subjects With New Onset of Autoimmune Diseases (NOADs)
Description: NOADs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: From Month 0 to Month 7.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 1 | 1 | 2 | 1

29. Secondary Outcome: Number of Subjects With New Onset of Autoimune Diseases (NOADs)
Description: NOADs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: From Month 0 to Month 48.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 3 | 4 | 5 | 4

30. Secondary Outcome: Number of Subjects With New Onset of Autoimmune Diseases (NOADs)
Description: NOADs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: Throughout the study period, from Month 0 to Month 60.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 4 | 4 | 5 | 6

31. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs)
Description: NOCDs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: From Month 0 to Month 7.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 4 | 2 | 6 | 3

32. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs)
Description: NOCDs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: From Month 0 to Month 48.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 8 | 11 | 13 | 6

33. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs)
Description: NOCDs include conditions such as autoimmune disorders, asthma, type I diabetes, or allergies.
Time Frame: Throughout the study period, from Month 0 to Month 60.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 8 | 11 | 14 | 7

34. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity, or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Month 0 to Month 7.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 4 | 4 | 4 | 2

35. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Month 0 to Month 48.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 10 | 13 | 19 | 13

36. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 35
Time Frame: Throughout the study period, from Month 0 to Month 60.
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Number analyzed (Participants) | 240 | 241 | 240 | 239
Participants | 14 | 16 | 19 | 15

ADVERSE EVENTS:
Time Frame: Serious adverse events: From Month 0 to Month 60. Unsolicited adverse events: Within the 30-day (Days 0-29) follow-up period after vaccination. Solicited symptoms: Within the 7-day (Days 0-6) follow-up period after vaccination.
Description: 3 among the serious adverse events (SAEs) listed below are SAEs reported for the subject's offsprings (Spina bifida, Foetal distress syndrome and Premature baby).
Arm/Group | Cervarix 1/Placebo Group | Cervarix 1/Placebo/Cervarix 1 Group | Cervarix 2/Placebo/Cervarix 2 Group | Cervarix 2 Group
Serious Adverse Events (participants affected / at risk) | 14/240 | 16/241 | 19/240 | 15/239
Other Adverse Events (participants affected / at risk) | 229/240 | 233/241 | 228/240 | 233/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix 1/Placebo Group (N=240) | Cervarix 1/Placebo/Cervarix 1 Group (N=241) | Cervarix 2/Placebo/Cervarix 2 Group (N=240) | Cervarix 2 Group (N=239)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Spina bifida (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 — SAE reported for the subject's offspring
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 4 | 1
Endometritis decidual (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 2
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Ligament laxity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basilar artery thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 — SAE reported for the subject's offspring
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 — SAE reported for the subject's offspring
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Anorexia nervosa (Psychiatric disorders) | 0 | 0 | 1 | 0
Bulimia nervosa (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix 1/Placebo Group (N=240) | Cervarix 1/Placebo/Cervarix 1 Group (N=241) | Cervarix 2/Placebo/Cervarix 2 Group (N=240) | Cervarix 2 Group (N=239)
Pain (General disorders) | 222 | 225 | 222 | 225
Redness (General disorders) | 109 | 112 | 123 | 145
Swelling (General disorders) | 92 | 88 | 83 | 118
Arthralgia (General disorders) | 45 | 57 | 39 | 43
Fatigue (General disorders) | 100 | 109 | 104 | 107
Fever (General disorders) | 23 | 20 | 22 | 39
Gastrointestinal (General disorders) | 48 | 48 | 36 | 68
Headache (General disorders) | 101 | 116 | 112 | 125
Myalgia (General disorders) | 79 | 109 | 98 | 99
Rash (General disorders) | 12 | 12 | 10 | 15
Nasopharyngitis (Infections and infestations) | 10 | 11 | 9 | 15

LIMITATIONS AND CAVEATS:
If appropriate, describe significant limitations of the trial. Examples: Early termination leading to small number of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.